CLINICAL TRIAL: NCT03558464
Title: Effectiveness of an Integrated Programme to Reduce Maternal and Child Malnutrition in Kenya: a Study in Pregnant Women and Their Offspring
Brief Title: Effectiveness Study During the First 1,000 Days in Kenya
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fabian Rohner (Other)
Collaborators: One Acre Fund (Unknown); Children's Investment Fund Foundation (Other)
Responsible Party: Sponsor-Investigator, Fabian Rohner, President, GroundWork
Organization: GroundWork (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GW_1AF_KenEff_1000d
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Stunting; Anemia; Micronutrient Deficiency
MeSH Terms: conditions — Growth Disorders; Anemia | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Cluster Randomized, Parallel-group, Prospective, Follow-up Effectiveness Study
Who Masked: Outcomes Assessor
Masking Description: The nature of the intervention package compared to the control package prevents a double-blind study design and thus, only the outcome assessors (data collectors) and the study statistician can be blinded to the group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Intervention (agriculture-focused package
  + nutrition-sensitive and nutrition-specific interventions=integrated package)
  Interventions: Dietary Supplement: Intervention (integrated package)
- Control (Active Comparator): (agriculture-focused package)
  Interventions: Other: Control

INTERVENTIONS:
Dietary Supplement: Intervention (integrated package) — During whole study (pregnant women and offspring):
  * Soap (for daily hand washing)
  * Chlorine solution (for daily drinking water treatment)
  * Life stage-appropriate (pregnancy, lactation, IYCF) monthly nutrition and WASH trainings
  During pregnancy and up to when offspring turns 6 months old:
  * LNS (Enov' Mum, 20g sachet daily)
  * Anthelminthic treatment (single-dose mebendazole (500mg), once during second trimester of pregnancy)
  Children 6-24 months of age
  * MNP (MixMe, 1g sachet every three days)
  * ORS + zinc
  * 1 egg per day
  All families in the intervention group will receive the same agriculture-focused package (see section 'control intervention' below) as those in the control group. All women will follow regular antenatal care as provided by the Kenyan government as part of their routine health system (e.g. intermittent preventive malaria treatment and iron-folic acid-supplements).
  Arms: Intervention
Other: Control — Active control: The families living in the control clusters will receive the agriculture-focused package that is already in place in all participating clusters through the 1AF programme. This agriculture focused package consists of: - Agricultural training (every 2 weeks on average) for all - Free to enrol for the following products on credit: o Compost boosters
  * Cook stoves o Seeds (onions, maize, indigenous greens, beans) o Maize storage bags o Drying tarps
  * Trees o Solar lights o Fertilizer o Actellic dust (insecticide) o Re-usable sanitary pads
  Arms: Control

SUMMARY:
Malnutrition is a public health problem in Kenya, with 26% of children underfive years of age stunted, and 26% of pre-school children, 26% of women of reproductive age and 42% of pregnant women being anaemic, respectively. Agriculture is the main source of income, food and nutrients for the majority of rural families in Sub-Saharan Africa including Kenya. Most farmers are smallholders and are vulnerable to poor nutrition. Thus far, programmes have mostly focused on increasing yields and household income, but not on improving nutritional status. One Acre Fund (1AF) has over the past 10 years successfully introduced an agriculture programme to smallholder farmers in Western Kenya focusing on improving harvest. 1AF is therefore well placed to transform an existing and successful agriculture programme into the world's largest 'nutrition network' for farmers, and it is the hope that a partnership between Children's Investment Fund Foundation (CIFF) and 1AF will create a strong voice for nutrition within the agriculture sector. The project aims to use an integrated programme by introducing nutrition-sensitive (improved water, sanitation and hygiene (WASH): e.g. soap for hand washing) and nutritionspecific (e.g. micronutrient supplements) components to 1AF's agricultural programme. The impact of such an integrated programme will be assessed in a cluster randomized intervention study in pregnant women and - after delivery - their offspring until they reach two years of age comparing one group receiving the integrated intervention to another group receiving the agricultural intervention (already in place).

DETAILED DESCRIPTION:
Background/Introduction

In partnership with the Children's Investment Fund Foundation (CIFF), 1AF aims to introduce nutrition-sensitive and nutrition-specific components into the services offered to smallholder farmer households. The nutrition-specific interventions consist of providing LNS to pregnant women up to 6 months after delivery and LNS to their offspring from 6-24 months of age. These nutritional supplements are recommended by WHO in areas where micronutrient deficiencies and malnutrition are prevalent. As a nutrition-sensitive intervention, pregnant women will receive mebendazole as preventive anthelminthic treatment after the first trimester.

In order to increase protein consumption, chicken birds will be provided to households. Further, children older than 6 months will be provided with oral rehydration salts (ORS) and zinc supplements as recommended by WHO and UNICEF for the treatment of acute diarrhoea [9]. Lastly, some WASH related interventions will also be provided, such as training sessions, soap for hand washing and chlorine for drinking water treatment.

To test the incorporation of nutrition services in 1AF's agricultural programme, pilot projects in western Kenya will be conducted between 2017 and 2020.

The dietary diversity, food frequency and subsequently, a minimum acceptably dietary quality for young children are lower in the Western Province than for the national average.

In order to monitor and evaluate 1AF's programmes, a cluster-randomized, parallel-group, prospective, follow-up effectiveness study that will span over the "1,000 days window", the period from conception until the child's second birthday will be conducted in the Western Province of Kenya.

Clusters will be randomly assigned to either have the regular 1AF agricultural intervention package (already in place in all clusters participating in the study and therefore called control) or the integrated intervention package that on top of the agricultural package consists of nutrition-specific (such as providing additional micronutrients) and nutrition-sensitive (such as providing soap for hand washing) interventions. The impact on malnutrition and programmatic 'success' will be evaluated.

Objective/hypothesis:

While the primary purpose is to longitudinally compare the changes of biological indicators such as growth, anemia and micronutrient status between the intervention and control group, the programmatic aspects such as adherence to and coverage of the intervention package and trying to link this to changes in dietary patterns and ultimately linear growth will also be evaluated.

As such, the research hypothesis is as follows: Linear growth in children during their first 24 months of life will improve after the provision of agricultural services, nutritionally enhanced and WASH products as well as nutrition and WASH training over the period of the 1,000 days window of opportunity when compared to the control group provided only with agricultural services.

Study design:

The general study design is a cluster-randomized, parallel-group, prospective, follow-up effectiveness study over a period of 1000 days comparing 2 groups:

1. Intervention group: Pregnant women will be given LNS (1 sachet/day) and an anthelminthic drug (mebendazole) in the second trimester of pregnancy, as well as soap and chlorine solution for the woman and the household. After delivery these products will be continued until the child reaches 6 months of age. Thereafter, LNS and anthelmintic drugs for mothers will be discontinued and instead, the child will receive MNP (1 sachet every three days), 1 egg per day, and Oral Rehydration Salts (ORS) along with zinc tablets (20 mg/day) for treatment in case of acute diarrhoea. These products will be given until the child reaches 2 years of age. The products will be accompanied by life stage-appropriate nutrition and WASH trainings (pregnancy, lactation, infant and young child feeding), as well as SMS reminders to highlight certain messages on antenatal care and nutrition. All products and trainings will be provided free of charge. The households in the intervention group will also have the same agricultural intervention as the control group.
2. Control group: All households will be provided with agricultural training (every 2 weeks on average) for free. In addition, households can also enrol for the following products on credit: compost booster, cook stoves, seeds (onions, maize, indigenous greens, beans), maize storage bags, drying tarps, trees, solar lights, fertilizer, actellic dust (insecticide), re-usable sanitary pads.

It is anticipated to enroll 1200 (600 in each group) pregnant women into the study; this is expected to yield a sufficiently large sample of children later in the study. Women will be recruited from 140 clusters (randomly assigned to intervention or control) that will be drawn from from Kimilili, Webuye, Bumula, Sirisia and Kabuchai districts in Bungoma County in Western Province of Kenya.

The communities will be informed about the study in village meetings by CHVs and by conducting outreach within their catchment area to identify pregnant women. Pregnant women will then be screened by 1AF enumerators. During screening, a few questions on health status and pregnancy will be asked. If the woman is prior or equal to 20 weeks of gestation (according to last menstrual period), has no visible severe disease and no allergy to peanuts or milk products, and confirms anticipated residence in the area for the coming 30 months, written informed consent for her and her offspring will be sought from her. She will then be asked to provide a urine sample to confirm pregnancy and she will be enrolled if pregnancy is confirmed. Following the screening, 5 assessment rounds (baseline and 4 follow-up assessments during the intervention) will be conducted at the participant's homes (rounds 1-3) or at a central place (rounds 4 and 5) within walking distance from their homes. Assessment round 3 (immediately) after delivery will be conducted as home visits or clinic visits in case of delivery at a clinic. Details of assessment procedures for each round are illustrated below:

Round 1 (Enrolment, ≤20 wk of gestation):

On the day of enrollment the round 1 assessment will be done. As part of this, the following information will be collected: household demographics and characteristics, maternal education; knowledge, attitude and practices (KAP) of specific dietary and nutrition practices during pregnancy; individual dietary diversity; antenatal care; WASH practices; height, weight and mid-upper arm circumference; maternal haemoglobin concentration and malaria parasitaemia from a capillary blood sample. After round 1, participants randomly allocated to the intervention group will start receiving the intervention package.

Round 2 (Gestational age of 34±1 wk):

In round 2, interview questions related to diet and nutrition KAP during pregnancy, dietary diversity, antenatal care, and WASH will be asked. Additionally, MUAC (mid-upper arm circumference) will be measured and a capillary blood sample for measurement of haemoglobin concentration, malaria parasitaemia and micronutrient status will be provided.

Round 3 (Within 24-48 hours after delivery):

The mother-child pair will be visited within 24-48 hours after delivery. The following information will be recorded: delivery date and time, delivery method, recent antenatal care, and early initiation of breastfeeding. The mother will be assessed for MUAC but no blood sampling will be conducted. For the newborn, head circumference, birth weight and birth length, and haemoglobin concentration (from a heelprick) will be measured.

Round 4 (At 6.5 mo ± 1 mo of age of offspring):

This assessment will be conducted when the child turns 6.5 months old. Breastfeeding and other infant and young child feeding indicators, child morbidity, maternal dietary diversity, postnatal care, and WASH information will be gathered. In mothers, MUAC and weight will be measured and haemoglobin concentration and malaria parasitaemia from a capillary sample will be assessed. In children, length, weight and head circumference will be measured and a capillary blood sample for haemoglobin concentration, malaria parasitaemia and micronutrient status will be provided.

Round 5 (At 24 ± 1mo of age of offspring):

This assessment will be conducted when the child turns 24 months old. Questionnaire-based information on child feeding, child dietary diversity, child morbidity and WASH will be collected. As in round 4, child length, weight and head circumference will be measured and a fingerprick blood sample will be provided for the measurement of haemoglobin concentration, malaria parasitaemia, and micronutrient status. No maternal biomarkers will be collected at this point.

As part of the monthly visits to the participants' households, the 1AF health field officers will also collect data on intervention adherence and recent morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women (≥ 18 years of age) with gestational age ≤20 weeks
* Written Informed Consent as documented by signature

Exclusion Criteria:

* Family does not intend to stay within the study area for at least the following 30 months
* Known history of allergy towards peanut or milk products
* Visible severe disease

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women will be enrolled (gender-specific) but for their offspring, inclusion is gender-independent
Enrollment: 1199 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Stunting and length/height-for-age z-score | 2 years
  Change in length-for-age z-score (LAZ) between birth and 24 months of age
Length-for-age z-score at 24 months of age | 24 months of age
  Update (October 2025): The outcome "Length-for-age z-score (LAZ) at 24 months of age" has been added to this record to correct an omission in the original registration. The trial's sample size calculation was based on this outcome (LAZ at 24 months), which was pre-specified as an outcome in the statistical analysis plan finalized before data analysis. The originally registered primary outcome, "change in LAZ between birth and 24 months," remains listed and is reported in the corresponding publication. This update represents a correction of a documentation error and does not constitute a post hoc change to the trial analysis.
  The length-for-age z-score (LAZ) is calculated using the WHO Child Growth Standards. It represents the number of standard deviations a child's length is from the median of healthy reference children of the same age and sex. Higher LAZ values indicate better linear growth. Typical biological ranges fall approximately between -6 and +6.

SECONDARY OUTCOMES:
Maternal hemoglobin | 8 months
  Change in haemoglobin concentration between 34 weeks gestation and 6 months post-partum
Birth weight | 7 months
  Differences in birth weight between intervention and control group
Birth length | 7 months
  Differences in birth length between intervention and control group
Head circumference at birth | 7 months
  Differences in head circumference between intervention and control group
Child hemoglobin | 2 years
  Change in hemoglobin concentration between at birth, 6 and 24 months of age
Child iron deficiency | 18 months
  Change in proportion with inflammation-adjusted iron deficiency between 6 and 24 months of age
Child vitamin A deficiency | 18 months
  Change in proportion with inflammation-adjusted vitamin A deficiency between 6 and 24 months of age
Child diarrhea | 18 months
  Diarrhea incidence rate between 6 and 24 months of age
Length-for-age z-score at birth and 6 months of age | At birth and 6 months of age
  Update (October 2025): This outcome was pre-specified in the data analysis plan (https://osf.io/rufmd) but was not originally listed in the ClinicalTrials.gov registration. This update reflects a correction of the registry to include the main planned secondary outcomes. This does not represent a post hoc addition to the initially planned statistical analyses (pre-specified in the data analysis plan).
  The length-for-age z-score (LAZ) is calculated using the WHO Child Growth Standards. It represents the number of standard deviations a child's length is from the median of healthy reference children of the same age and sex. Higher LAZ values indicate better linear growth. Typical biological ranges fall approximately between -6 and +6.
Proportion of stunted children (length-for-age z-score <-2 SD) at 6 and 24 months of age | At 6 months and 24 months of age
  Update (October 2025): This outcome was pre-specified in the data analysis plan (https://osf.io/rufmd) but was not originally listed in the ClinicalTrials.gov registration. This update reflects a correction of the registry to include the main planned secondary outcomes. This does not represent a post hoc addition to the initially planned statistical analyses (pre-specified in the data analysis plan).
  The length-for-age z-score (LAZ) is calculated using the WHO Child Growth Standards. It represents the number of standard deviations a child's length is from the median of healthy reference children of the same age and sex. Higher LAZ values indicate better linear growth. Typical biological ranges fall approximately between -6 and +6. A value below -2 SD is indicative for stunting and a value of below -3 SD for severe stunting.
Inflammation adjusted serum ferritin concentration at 6 and 24 months of age | At 6 and 24 months of age
  Update (October 2025): This outcome was pre-specified in the data analysis plan (https://osf.io/rufmd) but was not originally listed in the ClinicalTrials.gov registration. This update reflects a correction of the registry to include the main planned secondary outcomes. This does not represent a post hoc addition to the initially planned statistical analyses (pre-specified in the data analysis plan).
Retinol-binding protein at 6 and 24 months of age | At 6 and 24 months of age
  Update (October 2025): This outcome was pre-specified in the data analysis plan (https://osf.io/rufmd) but was not originally listed in the ClinicalTrials.gov registration. This update reflects a correction of the registry to include the main planned secondary outcomes. This does not represent a post hoc addition to the initially planned statistical analyses (pre-specified in the data analysis plan).

CONTACTS AND LOCATIONS:
Overall Officials: Rita Wegmüller, PhD, Principal Investigator — GroundWork
Locations (1):
- One Acre Fund, Kakamega, Kenya

IPD SHARING:
Plan to Share IPD: Undecided